CLINICAL TRIAL: NCT06174350
Title: Evaluation of the Effect of Cognitive Behavioral Therapy on Ruminative Thoughts and Cognitive Distortions in Individuals Exposed to Earthquakes
Brief Title: Evaluation of the Effect of Cognitive Behavioral Therapy in Individuals Exposed to Earthquakes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Adile Bozkurt Tonguc, Principal Investigator, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: OsmaniyeKAU-SBF-ABT-01
Record Dates: First submitted 2023-12-04; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Earthquake Victim
Keywords: Earthquakes; cognitive behavioral therapy; Rumination, Cognitive
MeSH Terms: conditions — Rumination Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: two groups: therapy group and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: There is a control and experimental group. Analysis was masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Cognitive behavioral therapy will be applied to the individuals in the experimental group who were exposed to the earthquake.
  Interventions: Behavioral: Cognitive behavioral therapy
- Placebo group (Experimental): No intervention will be applied to the control group of individuals exposed to the earthquake.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Earthquake is a process that affects the lives of many people. It is very important to evaluate the psychological state of individuals after the earthquake and take appropriate action. When studies conducted after the earthquake were examined, no study was found that evaluated the effect of cognitive behavioral therapy on ruminative thoughts and cognitive distortions in individuals exposed to earthquakes. For this reason, this thesis was conducted to evaluate the effect of cognitive behavioral therapy on ruminative thoughts and cognitive distortions in individuals exposed to earthquakes.
  Arms: experimental group
Other: Placebo — Intervention Description not
  Arms: Placebo group

SUMMARY:
Earthquake is a process that affects the lives of many people. It is very important to evaluate the psychological state of individuals after the earthquake and take appropriate action. When studies conducted after the earthquake were examined, no study was found that evaluated the effect of cognitive behavioral therapy on ruminative thoughts and cognitive distortions in individuals exposed to earthquakes. For this reason, this thesis was conducted to evaluate the effect of cognitive behavioral therapy on ruminative thoughts and cognitive distortions in individuals exposed to earthquakes.

DETAILED DESCRIPTION:
Earthquake is a process that affects the lives of many people. It is very important to evaluate the psychological state of individuals after the earthquake and take appropriate action. When studies conducted after the earthquake were examined, no study was found that evaluated the effect of cognitive behavioral therapy on ruminative thoughts and cognitive distortions in individuals exposed to earthquakes. For this reason, this thesis was conducted to evaluate the effect of cognitive behavioral therapy on ruminative thoughts and cognitive distortions in individuals exposed to earthquakes. In this thesis, a mixed design will be used in which quantitative and qualitative research methods will be used together.

* The quantitative dimension of the research will be carried out in an experimental design with pre-test, post-test control group and repeated measurement, and the qualitative dimension will be carried out with semi-structured questions that have a certain contact with individuals.
* The population of the research will be individuals in the container city in Osmaniye.
* The sample size will be determined by power analysis, and equal numbers of individuals will be included in the intervention and control groups.
* There will be 8-10 sessions for each individual, each session lasting 45-60 minutes.
* Sessions will be held between November 2023 and December 2023. The 3rd month follow-up will be done in March 2024.
* In this thesis, quantitative data, Socio-demographic Data Form, ruminative thought style scale and cognitive distortions scale will be used.
* Qualitative data were collected through semi-structured questions and therapy interviews.

will be collected.

* SPSS Statistics 20 program will be used in the analysis of qualitative data. MAXQDA Analytics Pro 2020 program will be used.
* Informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

being over 18 years old exposure to earthquake living in a container Ability to communicate

Exclusion Criteria:

Not being able to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Ruminative Thought Style Questionnaire (RTS) | 2 weeks
  İt was observed that internal consistency of the questionnaire were high (Cronbach alpha = 0.907). In the principal components and scree plot analysis revealed that the Turkish version of RTS has one component, and these explained %63.43 of total variance. In order to search for the convergent validity of RTS, the correlation between LESS-rumination sub-scale and The Metacognition Questionnaire was examined and meaningful relations were found. For the divergent validity, there appeared meaningful relation in a negative way, between the scores of RTS and LESS- Acceptance of Feelings and Comprehensibility sub-scales. Results: This study shows that Ruminative Thought Style Questionnaire can be used as a valid and reliable scale under Turkey conditions. The score that can be obtained from the scale varies between 20 and 140. There are no reverse items in the scale. The higher the score, the higher the rate of ruminative thoughts.

SECONDARY OUTCOMES:
THE COGNITIVE DISTORTIONS SCALE | 2 weeks
  Turkish and analyze its validity and reliability. Adapting the scale to Turkish, aimed at compliance with culture and the consequence of that in order to get more realistic results. In the scope of this study, different types of cognitive distortions and mental health variables were evaluated. There are no reverse items in the scale. Minimum 20 and maximum 140 points are received.

OTHER OUTCOMES:
qualitative questions | 2 weeks
  Qualitative questions about the earthquake and daily life will be asked and an evaluation will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Adile Bozkurt Tonguç, Principal Investigator — karaçay temporary accommodation center
Locations (1):
- Karaçay Temporary Accommodation Center, Osmaniye, Osmani̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No